CLINICAL TRIAL: NCT05175469
Title: Flow Cytometric Analysis of Peripheral Blood Neutrophil Myeloperoxidase Expression for Ruling Out Myelodysplastic Syndromes: Protocol for a Diagnostic Accuracy Study
Acronym: MPO-MDS-Valid
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC21.145; 2021-A01101-40 (Other: ID RCB)
Record Dates: First submitted 2021-12-14; First posted 2022-01-03 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Myelodysplastic Syndromes
Keywords: Myelodysplastic syndromes; Diagnostic accuracy study; Flow cytometry analysis; Myeloperoxidase; Peripheral blood sample; Additional relevant MeSH terms: Preleukemia, Syndrome, Disease, Pathologic Processes
MeSH Terms: conditions — Myelodysplastic Syndromes; Syndrome; Disease; Pathologic Processes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Flow cytometric analysis of neutrophil myeloperoxidase expression — Performance of flow cytometric analysis of neutrophil myeloperoxidase expression in peripheral blood samples will be blinded to the reference standard. Peripheral blood samples will be collected in 5 ml (EDTA) anticoagulant plastic tubes and processed on the same day of collection.
  Blood samples will be incubated with a panel of antibodies conjugated to fluorochromes, according to the manufacturers' recommendations.
  At least 10,000 cell events will be acquired on a 3-laser, 8/12-color flow cytometer and analyzed using flow cytometry software. Myeloperoxidase expression in the peripheral blood neutrophil population within an individual subject will be expressed as intra-individual robust coefficient of variation (RCV).

SUMMARY:
Myelodysplastic syndromes (MDS) are clonal bone marrow neoplasms characterized by dysplasia and ineffective hematopoiesis leading to peripheral blood cytopenias, with an increased risk of progression to acute myeloid leukemia. The conventional diagnostic work-up of MDS relies on cytomorphological evaluation of bone marrow, which may be complemented by conventional cytogenetic, flow cytometry, and molecular analysis by next generation sequencing techniques.

Suspicion of MDS is the commonest reason for bone marrow aspirate in older patients with unexplained peripheral blood cytopenias. Yet many patients are exposed to unnecessary bone marrow aspiration-related discomfort and harms, because of the limited prevalence of disease among subjects referred for suspected MDS. In this context, a valid and reliable assay based on peripheral blood sample that accurately discriminates MDS from other cytopenia etiologies without requiring invasive bone marrow aspiration is warranted.

The accuracy of peripheral blood neutrophil myeloperoxidase expression quantified by flow cytometric analysis for the diagnosis of MDS is supported by three primary studies totaling 211 individuals. An intra-individual robust coefficient of variation (RCV) value for neutrophil myeloperoxidase expression lower than 30.0% accurately ruled out MDS, with both sensitivity and negative predictive value point estimates of 100%, in consecutive patients with suspected disease. This biomarker might obviate the need for cytomorphological evaluation of bone marrow aspirate for up to 35% of patients referred for suspected MDS. Although promising, these preliminary results require replication in an independent external validation sample.

The broad aim of the multicenter MPO-MDS-Valid study project is to prospectively validate the diagnostic accuracy of intra-individual RCV for peripheral blood neutrophil myeloperoxidase expression quantified by flow cytometric analysis among consecutive patients referred for suspected MDS.

DETAILED DESCRIPTION:
The primary objective of the MPO-MDS-Valid study is to estimate the discriminative accuracy (i.e., area under the ROC curve point estimate along with 95% confidence interval [CI]) of the intra-individual RCV for neutrophil myeloperoxidase expression in peripheral blood for the diagnosis of MDS in consecutive patients.

The secondary objectives are:

1. To estimate the negative predictive value of the intra-individual RCV for neutrophil myeloperoxidase expression in peripheral blood (with a prespecified threshold of 30.0%) for ruling out MDS in consecutive patients.
2. To estimate the prevalence of alternate diagnoses established by bone marrow cytomorphology among true negative patients (i.e., patients with intra-individual RCV value lower than 30.0% and for whom MDS was ruled out by the reference method).

Study design: The MPO-MDS-Valid study project is a multicenter diagnostic accuracy study of an index test by comparison with a reference standard in unselected consecutive patients. An institutional review board (Comité de Protection des Personnes Nord Ouest III) reviewed and approved the study protocol and the information form, prior to study initiation. No specific intervention is assigned to participants. All diagnostic testing, procedures, and medication ordering are performed at the discretion of attending physicians. The index test result will have no impact on patient management.

Screening: All consecutive patients referred for suspicion of MDS to the immuno-hematology lab at the study sites will be screened for eligibility. A lab physician will review inclusion and exclusion criteria, using computerized medical and laboratory records.

Recruitment: Participants will be included in the study once all the screening activities have been conducted and only if the patient meets all inclusion and none exclusion criteria. The consent for flow cytometry analysis of peripheral blood sample and data collection through chart review will be sought under a regime of "non-opposition" (opt-out): after appropriate written information is delivered, data will be collected except in case of opposition from the patient. All patients included in the study will be assigned a unique patient identification number. This number will be used to identify the patient throughout the study.

Index test: Flow cytometric analysis of neutrophil myeloperoxidase expression in peripheral blood will be blinded to the reference standard. Myeloperoxidase expression in the peripheral blood neutrophil population within an individual subject will be expressed as RCV. The intra-individual RCV is calculated as the robust standard deviation divided by the median. The robust standard deviation is a function of the deviation of individual data points to the median of the study population. Intra-individual RCV is expressed as percentage and reflects the variability in myeloperoxidase expression in the peripheral blood neutrophil population within an individual subject.

Reference standard: At each study site, cytomorphological evaluation of bone marrow aspirate will be performed by experienced hematopathologists blinded to the index test.

Morphologic assessment may be complemented by bone marrow flow cytometric score, karyotype, and molecular profiling, where relevant. The reference criteria for MDS are 1) the presence of ≥10% dysplastic cells in any hematopoietic lineage on bone marrow aspirate, and 2) the exclusion of acute myeloid leukemia (defined by the presence of ≥20% bone marrow blasts). Consistent with WHO classification, MDS subcategorization will be based on the degree of dysplasia (unilineage versus multilineage), blast percentages, presence of ring sideroblasts, and cytogenetic analysis (del(5q)).

The reference criteria for chronic myelomonocytic leukemia (CMML) diagnosis are 1) the presence of persistent peripheral blood monocytosis ≥1 x109/L, and 2) monocyte accounting for more than 10% of the white blood cell differential count. Idiopathic cytopenia of uncertain significance (ICUS) will be defined by unexplained mild persistent cytopenia for 4 to 6 months and the failure to establish the diagnosis of MDS according to reference criteria.

Patients with confirmed suspicion of MDS: Participants for whom the diagnosis of MDS (or CMML) is confirmed by the reference standard will be categorized as patients with confirmed suspicion of MDS.

Patients with unconfirmed suspicion of MDS: Participants for whom the diagnosis of MDS (or CMML) is ruled out by the reference standard will be categorized as patients with unconfirmed suspicion of MDS. This latter subgroup will include patients with ICUS, as defined in accordance with published guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Age at enrollment ≥18 years
* Referral for suspicion of myelodysplastic syndrome
* Indication for bone marrow examination
* ≥1 peripheral blood cytopenia defined by hemoglobin concentration <12 g/dL for female and <13g/dL for male patients, platelet count <150 x109/L, absolute neutrophil count <1.8 x109/L
* Inpatient or outpatient care

Exclusion Criteria:

* Refusal to participate
* History of or active documented MDS or CMML
* Enrollment in intensive or critical care unit
* Incarcerated or individuals protected by French regulation (Article L1121.5 and following, Code de la Santé Publique)
* Not affiliated with social security system
* Previous enrollment in the study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult, Older Adult
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Area under the receiver operating characteristic (ROC) curve | Baseline
  The area under the ROC curve point estimate along with 95% confidence interval will quantify the accuracy of the index test (i.e., intra-individual RCV for neutrophil myeloperoxidase expression in peripheral blood) for the diagnosis of myelodysplastic syndromes (MDS) or chronic myelomonocytic leukemia (CMML). The reference diagnosis will be established by cytomorphological evaluation of bone marrow aspirate performed by independent experienced hematopathologists blinded to the index test results. Morphologic assessment may be complemented by bone marrow flow cytometric score, karyotype, and molecular profiling, where relevant.

SECONDARY OUTCOMES:
Negative predictive value | Baseline
  The negative predictive value point estimate along with 95% confidence interval for the index test (i.e., intra-individual robust coefficient of variation with a prespecified threshold of 30.0%) will be computed by comparison with the reference standard for myelodysplastic syndromes (MDS) or chronic myelomonocytic leukemia (CMML)
Prevalence of alternate diagnoses for true negative cases | Baseline
  Prevalence point estimate (along with 95% confidence interval) of alternate diagnosis established by bone marrow examination for unconfirmed suspicions of myelodysplastic syndromes with intra-individual RCV< 30.0% for neutrophil myeloperoxidase expression in peripheral blood.

CONTACTS AND LOCATIONS:
Overall Officials: Tatiana RASKOVALOVA, Principal Investigator — University Hospital, Grenoble
Locations (8):
- France (8):
  - University Hospital, Clermont-Ferrand, Clermont-Ferrand
  - Grenoble_Alpes UniversityHospital, Grenoble
  - University Hospital Lyon Sud, HCL, Lyon
  - Institut Paoli Calmettes, Marseille
  - University Hospital Saint-Eloi, Montpellier
  - Chu Nantes, Nantes
  - University Hospital NICE, Nice
  - University Hospital, Saint-Étienne, Saint-Etienne

IPD SHARING:
Plan to Share IPD: Yes
The principal investigator will respond directly to data requests by providing a de-identified data set. Individual participant data that underlie the results reported in the published articles (i.e., main text, tables, figures, and appendices) will be supplied.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 24 months after publication of the main findings of the final dataset.
  No end date.
Access Criteria: De-identified data will be available for individual participant data meta-analysis purpose.
  Researchers should submit a methodologically sound proposal that complies with the Preferred Reporting Items for Systematic Review and Meta-Analysis Protocols (PRISMA-P) 2015 statement. Proposals should be directed to TRaskovalova@chu-grenoble.fr. Data requestors will need to sign a data access agreement.

REFERENCES:
- [Derived] Planta C, Bret C, Manzoni D, Lhoumeau AC, Mayeur Rousse C, Ticchioni M, Campos L, Eischen A, Gonnet N, Merle R, Seigneurin A, Paul F, Comte E, Allieri-Rosenthal A, Tondeur S, Regnart C, Jacob MC, Labarere J, Park S, Raskovalova T. Flow cytometric analysis of peripheral blood neutrophil myeloperoxidase expression in myelodysplastic neoplasms (MPO-MDS-Valid): protocol for a multicentre diagnostic accuracy study. BMJ Open. 2024 Jun 17;14(6):e081200. doi: 10.1136/bmjopen-2023-081200. PMID 38889946